CLINICAL TRIAL: NCT01020253
Title: A Comparison of Alendronate vs. Alfacalcidol Medication for the Preservation of Bone Mineral Density Around the Femoral Implant and in the Lumbar Spine After a Total Hip Arthroplasty
Brief Title: The Effectiveness of Two Osteoporosis Drugs on Prosthetic Bone Mineral Density (BMD) Loss After Total Hip Arthroplasty(THA)
Acronym: ETOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Naoyuki Iwamoto, Yokohama City University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YCU07-122
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Bone Density; Arthroplasty, Replacement, Hip
Keywords: bisphosphonate, vitamin D3; Total Hip arthroplasty
MeSH Terms: interventions — Alendronate; alfacalcidol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alendronate medication (Active Comparator)
  Interventions: Drug: alendronate, alfacalcidol
- Alfacalcidol medication (Active Comparator)
  Interventions: Drug: alendronate, alfacalcidol
- Non-medication (No Intervention)
  Interventions: Drug: alendronate, alfacalcidol

INTERVENTIONS:
Drug: alendronate, alfacalcidol — Alendronate: 5mg per day, Tablet, Duration is 48 weeks. Alfacalcidol: 1μg per day, Tablet, Duration is 48 weeks.

SUMMARY:
The purpose of this study is to evaluate whether alendronate and alfacalcidol are effective on prosthetic or lumbar spine BMD after total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the hip
* patients after total hip arthroplasty

Exclusion Criteria:

* diseases related to bone metabolism
* patients taking drugs which affect bone metabolism

Ages: 44 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
DEXA QDR 2000, Hologic Co. | 1, 12, 24 and 48 weeks after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of orthopaedic surgery, Yokohama City University, Yokohama, Kanagawa, Japan